CLINICAL TRIAL: NCT05694169
Title: A Phase 1, Open-label, Supplemental Dosing Study of Participants With Chronic Kidney Disease Previously Treated With REACT (REGEN-015)
Brief Title: A Study of Participants With Chronic Kidney Disease Previously Treated With REACT
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: business decision
Sponsor: Prokidney (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REGEN-015
Record Dates: First submitted 2022-12-27; First posted 2023-01-23 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Diabetic Kidney Disease; CAKUT; Chronic Kidney Diseases
Keywords: REACT; CAKUT; DKD
MeSH Terms: conditions — Diabetic Nephropathies; Cakut; Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Renal Autologous Cell Therapy (REACT) (Experimental): Participants will receive 2 REACT injections separated by 6 months. All participants will be followed for 12 months post last supplemental REACT injection.
  Interventions: Biological: Renal Autologous Cell Therapy (REACT)

INTERVENTIONS:
Biological: Renal Autologous Cell Therapy (REACT) — Autologous selected renal cells (SRC)

SUMMARY:
The purpose of this study is to evaluate the safety of supplemental REACT injections in participants with chronic kidney disease (CKD) who have previously received REACT treatment.

DETAILED DESCRIPTION:
A Phase 1, Open-label trial where up to 10 participants will enroll in the trial after parent REACT protocol EOS visit completion. Participants may undergo a biopsy to manufacture REACT if additional biopsy tissue is required. Participants will receive 2 REACT injections separated by 6 months. All participants will be followed for 12 months post last supplemental REACT injection.

ELIGIBILITY:
Inclusion Criteria:

1. The participant has received REACT in a previous trial for treatment of chronic kidney disease and completed their parent protocol follow up period.
2. The participant is male or female, 30 to 80 years of age on the date of informed consent.
3. The participant has a documented clinical diagnosis of an eGFR greater than or equal to 14 and less than or equal to 50 mL/min/1.73m2, not requiring renal dialysis.
4. The participant has stable blood pressure and is maintained on a stable antihypertensive medication regimen if treatment for hypertension is necessary.

Exclusion Criteria:

1. The participant has a history of renal transplantation.
2. The participant has received dialysis for more than 30 days.
3. The participant has received any other investigational products after completion of REACT injections within 3 months of screening.
4. The participant has a urinary albumin-to-creatinine ratio (UACR) of greater than 5,000 mg/g.
5. The participant has hemoglobin levels less than 10 g/dL and is not responsive to the standard medical intervention for CKD-related anemia prior to screening.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2023-07-11 (Actual); Primary Completion 2024-03-19 (Actual); Study Completion 2024-05-13 (Actual)

PRIMARY OUTCOMES:
Primary Endpoints is as follows: | through 12 months after last supplemental injection
  Procedure and investigational product-related treatment-emergent adverse events (TEAE) will be assessed via:
  1. Biopsy Related SAEs
  2. Injection Procedure Related SAEs
  3. Investigational Product Related SAEs
  4. Treatment-Emergent SAEs.

SECONDARY OUTCOMES:
First Secondary Endpoint | 12 months after the last supplemental injection
  Percent of participants who have the same or reduced 5-year risk of end stage renal disease (ESRD)
Second Secondary Endpoint | 12 months after the last supplemental injection
  Percent of participants who have the same or reduced 2-year risk of ESRD

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Prokidney
Locations (1):
- Boise kidney and Hypertension Institute, Boise, Idaho, United States